CLINICAL TRIAL: NCT01290952
Title: ON Pump vs OFF Pump Myocardial Revascularization in High Risk Patients: a Randomized Study
Brief Title: On Versus Off Pump Myocardial Revascularization Study
Acronym: On-Off
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Italia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030211
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease
Keywords: off-pump; bypass; coronary artery surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Off-pump bypass surgery (Experimental): Off-pump coronary artery bypass graft (OPCAB) using mandatory a stabilization device and advisable, but not mandatory, a heart positioner
  Interventions: Procedure: Off-pump bypass surgery
- On-pump bypass surgery (Active Comparator): coronary artery bypass graft with cardiopulmonary bypass (CPB/CAB)
  Interventions: Procedure: On-pump bypass surgery

INTERVENTIONS:
Procedure: Off-pump bypass surgery — is a method of performing a coronary bypass operation for the purpose of treating advanced coronary heart disease while the heart is still beating normally.
  Arms: Off-pump bypass surgery
Procedure: On-pump bypass surgery — is a technique that temporarily takes over the function of the heart and lungs during surgery, maintaining the circulation of blood and the oxygen content of the body.
  Arms: On-pump bypass surgery

SUMMARY:
Compare completeness and modality of revascularization, operative and postoperative results and 1 year clinical outcomes in unselected high risk patients referred for primary coronary artery bypass surgery. Patients will be randomized to undergo off-pump coronary artery bypass graft (OPCAB) or coronary artery bypass graft with cardiopulmonary bypass (CPB/CAB).

DETAILED DESCRIPTION:
The initial application of off-pump coronary artery bypass in the early nineties was mainly directed to highly selected and relatively low risk surgical patients. Since then there has been a growing body of evidence suggesting many potential advantages of the OPCAB technique over the conventional cardiopulmonary bypass (CPB) technique in different groups of high-risk patients.

On-off study is a multicentre, prospective, randomized, parallel, trial.Patients indicated for elective or urgent isolated coronary artery bypass graft with additive European System for Cardiac Operative Risk Evaluation ≥ 6 were enrolled. Patients in cardiogenic shock were excluded. Patients were randomly assigned either to coronary artery bypass surgery with cardiopulmonary bypass (ON arm) or to off-pump coronary artery bypass graft (OFF arm). The composite primary end point included operative mortality, myocardial infarction, stroke, renal failure, re-operation for bleeding and adult respiratory distress syndrome, within 30 days after surgery. The total planned sample size was 693 patients; the actual number of enrolled patients was 411,according to the results of the interim analysis scheduled at 400 enrollments (alfa-spending=0.029, Pocock method).

ELIGIBILITY:
Inclusion Criteria:

* Pts candidate to a myocardial revascularization for any patter of coronary artery disease, ventricular dysfunction or any other co-morbidity
* EUROSCORE ≥ 6
* Pts who signed the Informed Consent
* Age ≥ 18 years

Exclusion Criteria:

* Patients in cardiogenic shock requiring emergency surgery or preoperative intra-aortic balloon pump
* Patients requiring additional surgical procedures
* Porcelain Aorta
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Lemma, Dr., Principal Investigator — Ospedale Sacco-Milano
Locations (8):
- Italy (7):
  - Policlinico, Bari
  - S. Anna e S. Sebastiano, Caserta
  - Ospedale Luigi Sacco, Milan
  - European Hospital, Roma
  - Ospedale S. Camillo, Roma
  - Ospedale S. Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale Molinette, Torino
- University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The main manuscript with the results of the primary endpoint analysis was published in December 2011.There are no plans to make individual partecipant data available

REFERENCES:
- [Background] Benetti FJ, Naselli G, Wood M, Geffner L. Direct myocardial revascularization without extracorporeal circulation. Experience in 700 patients. Chest. 1991 Aug;100(2):312-6. doi: 10.1378/chest.100.2.312. PMID 1677884
- [Background] Yokoyama T, Baumgartner FJ, Gheissari A, Capouya ER, Panagiotides GP, Declusin RJ. Off-pump versus on-pump coronary bypass in high-risk subgroups. Ann Thorac Surg. 2000 Nov;70(5):1546-50. doi: 10.1016/s0003-4975(00)01922-6. PMID 11093485
- [Background] Arom KV, Flavin TF, Emery RW, Kshettry VR, Janey PA, Petersen RJ. Safety and efficacy of off-pump coronary artery bypass grafting. Ann Thorac Surg. 2000 Mar;69(3):704-10. doi: 10.1016/s0003-4975(99)01510-6. PMID 10750747
- [Background] D'Ancona G, Karamanoukian HL, Soltoski P, Salerno TA, Bergsland J. Changing referral pattern in off-pump coronary artery bypass surgery: a strategy for improving surgical results. Heart Surg Forum. 1999;2(3):246-9. PMID 11276485
- [Background] Ascione R, Lloyd CT, Gomes WJ, Caputo M, Bryan AJ, Angelini GD. Beating versus arrested heart revascularization: evaluation of myocardial function in a prospective randomized study. Eur J Cardiothorac Surg. 1999 May;15(5):685-90. doi: 10.1016/s1010-7940(99)00072-x. PMID 10386418
- [Background] Vallely MP, Bannon PG, Kritharides L. The systemic inflammatory response syndrome and off-pump cardiac surgery. Heart Surg Forum. 2001;4 Suppl 1:S7-S13. No abstract available. PMID 11178301
- [Background] Cartier R, Brann S, Dagenais F, Martineau R, Couturier A. Systematic off-pump coronary artery revascularization in multivessel disease: experience of three hundred cases. J Thorac Cardiovasc Surg. 2000 Feb;119(2):221-9. doi: 10.1016/S0022-5223(00)70176-0. PMID 10649196
- [Background] Krejca M, Skiba J, Szmagala P, Gburek T, Bochenek A. Cardiac troponin T release during coronary surgery using intermittent cross-clamp with fibrillation, on-pump and off-pump beating heart. Eur J Cardiothorac Surg. 1999 Sep;16(3):337-41. doi: 10.1016/s1010-7940(99)00234-1. PMID 10554854
- [Background] Ascione R, Nason G, Al-Ruzzeh S, Ko C, Ciulli F, Angelini GD. Coronary revascularization with or without cardiopulmonary bypass in patients with preoperative nondialysis-dependent renal insufficiency. Ann Thorac Surg. 2001 Dec;72(6):2020-5. doi: 10.1016/s0003-4975(01)03250-7. PMID 11789787
- [Background] Kilo J, Czerny M, Gorlitzer M, Zimpfer D, Baumer H, Wolner E, Grimm M. Cardiopulmonary bypass affects cognitive brain function after coronary artery bypass grafting. Ann Thorac Surg. 2001 Dec;72(6):1926-32. doi: 10.1016/s0003-4975(01)03199-x. PMID 11789773
- [Background] Calafiore AM, Di Mauro M, Contini M, Di Giammarco G, Pano M, Vitolla G, Bivona A, Carella R, D'Alessandro S. Myocardial revascularization with and without cardiopulmonary bypass in multivessel disease: impact of the strategy on early outcome. Ann Thorac Surg. 2001 Aug;72(2):456-62; discussion 462-3. doi: 10.1016/s0003-4975(01)02810-7. PMID 11515882
- [Background] Al-Ruzzeh S, Nakamura K, Athanasiou T, Modine T, George S, Yacoub M, Ilsley C, Amrani M. Does off-pump coronary artery bypass (OPCAB) surgery improve the outcome in high-risk patients?: a comparative study of 1398 high-risk patients. Eur J Cardiothorac Surg. 2003 Jan;23(1):50-5. doi: 10.1016/s1010-7940(02)00654-1. PMID 12493504
- [Background] Vlassov GP, Deyneka CS, Travine NO, Timerbaev VH, Ermolov AS. Acute myocardial infarction: OPCAB is an alternative approach for treatment. Heart Surg Forum. 2001;4(2):147-50; discussion 150-1. PMID 11544627
- [Background] Yeatman M, Caputo M, Ascione R, Ciulli F, Angelini GD. Off-pump coronary artery bypass surgery for critical left main stem disease: safety, efficacy and outcome. Eur J Cardiothorac Surg. 2001 Mar;19(3):239-44. doi: 10.1016/s1010-7940(01)00572-3. PMID 11251259
- [Background] Geissler HJ, Holzl P, Marohl S, Kuhn-Regnier F, Mehlhorn U, Sudkamp M, de Vivie ER. Risk stratification in heart surgery: comparison of six score systems. Eur J Cardiothorac Surg. 2000 Apr;17(4):400-6. doi: 10.1016/s1010-7940(00)00385-7. PMID 10773562
- [Background] Nashef SA, Roques F, Michel P, Gauducheau E, Lemeshow S, Salamon R. European system for cardiac operative risk evaluation (EuroSCORE). Eur J Cardiothorac Surg. 1999 Jul;16(1):9-13. doi: 10.1016/s1010-7940(99)00134-7. PMID 10456395
- [Background] Shroyer AL, Grover FL, Hattler B, Collins JF, McDonald GO, Kozora E, Lucke JC, Baltz JH, Novitzky D; Veterans Affairs Randomized On/Off Bypass (ROOBY) Study Group. On-pump versus off-pump coronary-artery bypass surgery. N Engl J Med. 2009 Nov 5;361(19):1827-37. doi: 10.1056/NEJMoa0902905. PMID 19890125
- [Background] Khan NE, De Souza A, Mister R, Flather M, Clague J, Davies S, Collins P, Wang D, Sigwart U, Pepper J. A randomized comparison of off-pump and on-pump multivessel coronary-artery bypass surgery. N Engl J Med. 2004 Jan 1;350(1):21-8. doi: 10.1056/NEJMoa031282. PMID 14702424
- [Background] Puskas JD, Thourani VH, Kilgo P, Cooper W, Vassiliades T, Vega JD, Morris C, Chen E, Schmotzer BJ, Guyton RA, Lattouf OM. Off-pump coronary artery bypass disproportionately benefits high-risk patients. Ann Thorac Surg. 2009 Oct;88(4):1142-7. doi: 10.1016/j.athoracsur.2009.04.135. PMID 19766798

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 630 patients was the planned estimated sample size needed to test the null hypothesis. An interim analysis was scheduled at 400 enrolled patients, to verify the null hypothesis used for the sample size calculation. A p<0.0294 was considered statistically significant to reject the null hypothesis, thus study enrollment was stopped at 411 patients.
Groups:
- Off Pump: Off-pump coronary artery bypass graft (OPCAB) using mandatory a stabilization device and advisable, but not mandatory, a heart positioner
  Off-pump bypass surgery: is a method of performing a coronary bypass operation for the purpose of treating advanced coronary heart disease while the heart is still beating normally.
- On-pump: coronary artery bypass graft with cardiopulmonary bypass (CPB/CAB)
  On-pump bypass surgery: is a technique that temporarily takes over the function of the heart and lungs during surgery, maintaining the circulation of blood and the oxygen content of the body.
Period: Overall Study
Arm/Group | Off Pump | On-pump
Started | 204 | 207
Completed | 192 | 193
Not Completed | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Off Pump | On-pump | Total
Number analyzed (Participants) | 204 | 207 | 411
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 204 | 207 | 411
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 67 | 126
  Male | 145 | 140 | 285
Region of Enrollment [Number; unit: participants]
  Italy | 189 | 196 | 385
  Switzerland | 15 | 11 | 26
Euroscore > 6 (high risk for early mortality for cardiac surgery) [Number; unit: participants] | 204 | 207 | 411

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Post-operative Combined Endpoint (i.e. With One or More of the Following)
Description: Number of patients with one or more of the following:
  * Operative Mortality
  * Myocardial Infarction
  * Postoperative neurological complications
  * Renal failure
  * ARDS (Acute Respiratory Distress Syndrome)
  * Bleeding
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Off Pump | On-pump
Number analyzed (Participants) | 204 | 207
participants | 13 | 26

2. Secondary Outcome: Number of Patients With Secondary Combined Endpoint (i.e. With One or More of the Following)
Description: Number of patients with one of more of the following:
  * Post-operative Atrial Fibrillation
  * IAPB (Intra-Aortic Balloon Pump) insertion and low cardiac output syndrome
  * Ventilation > 24h
  * Sternal wound infection or dehiscence
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | On-pump Bypass Surgery | Off-pump Bypass Surgery
Number analyzed (Participants) | 207 | 204
participants | 73 | 67

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Off Pump | On-pump
Serious Adverse Events (participants affected / at risk) | 16/204 | 30/207
Other Adverse Events (participants affected / at risk) | 72/204 | 79/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off Pump (N=204) | On-pump (N=207)
Overall mortality (Cardiac disorders) | 12 (12) | 14 (14)
MACE (Cardiac disorders) | 4 (4) | 16 (16)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off Pump (N=204) | On-pump (N=207)
angina (Cardiac disorders) | 5 (5) | 6 (6)
Post-operative AF (Cardiac disorders) | 44 (44) | 44 (44)
IABP insertion (Cardiac disorders) | 7 (7) | 4 (4) — Intra Aortic Balloon Pump Insertion
Ventilation >24 h (Injury, poisoning and procedural complications) | 9 (9) | 15 (15)
Wound infection (Injury, poisoning and procedural complications) | 7 (7) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No